CLINICAL TRIAL: NCT00584454
Title: Continued Evaluation of the Safety of Q Fever Vaccine, Phase I, Inactivated, Freeze Dried, NDBR 105, in Those at Risk of Exposure to Coxiella Burnetii, A Phase 2 Study
Brief Title: Safety Evaluation of a Q-fever Vaccine, NDBR 105
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-13480; FY05-14 (Other: USAMRIID)
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Q Fever
Keywords: Coxiella burnetti, Bacterial Infections, Rickettsia, Hepatits, Endocarditis
MeSH Terms: conditions — Q Fever; Bacterial Infections; Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Q Fever Vaccine (NDBR 105) (Experimental): Volunteers will receive and intradermal dose of 0.1 ml of the skin test antigen (Q fever Skin Test Antigen, Henzerling Strain, Phase 1, MNLBR 110) in the volar aspect of the arm. Skin test will be evaluated; if erythema occurs after the skin test, it is medically contraindicated to vaccinate that volunteer. Volunteers with skin test reactions will not be vaccinated and withdrawn from the study.
  Interventions: Biological: Q Fever Vaccine (NDBR 105

INTERVENTIONS:
Biological: Q Fever Vaccine (NDBR 105 — Each volunteer will receive an intradermal dose of 0.1 ml of the skin test antigen (Q fever Skin Test Antigen, Henzerling Strain, Phase I, MNLBR 110) in the volar aspect of the arm on Day -7 of the study.Volunteers with skin test reactions that are considered negative may be vaccinated with Q Fever Vaccine, Phase I, Inactivated, Freeze-Dried, NDBR 105 (subcutaneously, 0.5 ml) in the upper outer aspect of the arm on Day 0 of the study.

SUMMARY:
The purpose of this study is to evaluate the safety of Q Fever vaccine, NDBR 105, and collect data on incidence of occupational Q Fever infection in at risk personnel.

DETAILED DESCRIPTION:
Study Objectives:

1. Continue to collect and assess safety data on Q Fever Vaccine, Phase I, Inactivated, Freeze-Dried, NDBR 105, and 2) Provide vaccine that potentially protects personnel at risk for occupational exposure to Q Fever and collect data on incidence of occupational Q Fever infection (subclinical and clinical) in immunized personnel.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old, or if on active military duty, 17 years old.
* Females of childbearing potential must agree to have a urine pregnancy test on the same day before receipt of skin test antigen AND vaccine. (Exception: documented hysterectomy or > three years of menopause.) The results must be negative.
* Volunteer must be actively enrolled in the SIP
* Volunteer must be considered at risk for exposure to C. burnetii.
* Volunteer must sign and date the approved ICD and HIPAA Authorization.
* Volunteer must have an up-to-date (within one year) medical history, physical examination, and laboratory tests on their charts and be medically cleared for participation by an Investigator. Examinations or tests may be repeated within one year at the discretion of the enrolling physician.
* Volunteer must be willing to return for all follow-up visits.
* Volunteer must agree to report any AEs which may or may not be associated with administration of the test article for at least 28 days after vaccination. All SAEs and UAEs will be reported for the duration of the volunteer's participation in the study (one year).

Exclusion Criteria:

* Prior history of Q fever disease or vaccination.
* Clinically significant abnormal lab results including evidence of Hepatitis C, Hepatitis B carrier state, or elevated liver function tests (two times the normal range or at the discretion of the PI).
* Personal history of an immunodeficiency or current treatment with an immunosuppressive medication or autoimmune disease.
* Confirmed HIV infection.
* Heart valve disease: murmur with abnormal echocardiogram (if murmur is detected on examination, volunteer will be referred to cardiologist to rule out pathology.)
* Positive pregnancy test or lactating female (females must agree to not become pregnant for three months after vaccination.)
* Any known allergies to components of the vaccine.
* Administration of another inactivated vaccine within 7 days or a live or IND vaccine within 28 days of Q fever vaccination.
* Any unresolved AE resulting from a previous immunization.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02; Primary Completion 2009-07 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Goldberg, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subject with negative skin test antigen were enrolled in this study
Pre-assignment Details: Patients were excluded from this study if after the skin test antigen erythema (> 30mm) or induration (> 20 mm) occured
Groups:
- Q Fever Vaccine (NDBR 105): Volunteers will receive and intradermal dose of 0.1 ml of the skin test antigen (Q fever Skin Test Antigen, Henzerling Strain, Phase 1, MNLBR 110) in the volar aspect of the arm. Skin test will be evaluated; if erythema occurs after the skin test, it is medically contraindicated to vaccinate that volunteer. Volunteers with skin test reactions will not be vaccinated and withdrawn from the study.
  Q-Fever Vaccine, NDBR 105: Each volunteer will receive an intradermal dose of 0.1 ml of the skin test antigen (Q fever Skin Test Antigen, Henzerling Strain, Phase I, MNLBR 110) in the volar aspect of the arm on Day -7 of the study.Volunteers with skin test reactions that are considered negative may be vaccinated with Q Fever Vaccine, Phase I, Inactivated, Freeze-Dried, NDBR 105 (subcutaneously, 0.5 ml) in the upper outer aspect of the arm on Day 0 of the study.
Period: Overall Study
Arm/Group | Q Fever Vaccine (NDBR 105)
Started | 10
Completed | 6
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Relocation | 1
Not completed — Clinical Hold | 2

BASELINE CHARACTERISTICS:
Arm/Group | Q Fever Vaccine (NDBR 105)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Adverse Reaction and Occupational Illness Endpoint Measurements in This Q Fever NDBR 105 Vaccine Study Will be Evaluated for All Intent-to-treat Volunteers.
Description: Observe adverse reactions and occupational illness endpoint measurements 7 days follow-up after receipt of skin test antigen and 12 months of follow-up after receipt of vaccine
Time Frame: AEs recorded through day 28 after vaccination; SAEs recorded through duration of study; Confirmed occupational illness recorded through duration of study
Population: Subjects at risk of exposure to Coxiella Burnetti (Q Fever)
Measure: Count of Participants; unit: Participants
Arm/Group | Q Fever Vaccine (NDBR 105)
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Q Fever Vaccine (NDBR 105)
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q Fever Vaccine (NDBR 105) (N=10)
Chills (General disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q Fever Vaccine (NDBR 105) (N=10)
Injection Site Erythema (General disorders) | 1 (1)
Injection Site Haematoma (General disorders) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site induration (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Injection site warmth (General disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Thirst (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No